CLINICAL TRIAL: NCT02726230
Title: Bihar Family Health Initiative (Ananya)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Anita Raj, Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BMGF#22539
Record Dates: First submitted 2016-03-21; First posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Maternal and Child Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ananya Intervention (Experimental): 1. Strengthen enumeration and mapping of areas to ensure reach of front line workers (FLWs: auxiliary nurse midwives- ANMs; community health workers- ASHAs; anganwadi workers- AWWs).
  2. Convene monthly FLW meetings to build skills and get trained in job kits to increase the quantity and quality of household visits.
  3. Train FLWs on communication skills and use of mobile kunji, a job-aid tool, to improve FLWs' communication with households.
  4. A mass media campaign inclusive of street theatre, tv and radio, and a mobile van.
  5. Community mobilization linking mass media efforts with self-help groups.
  6. Quality improvement activities at public health facilities.
  7. Facility-based skills training to staff delivering infants to improve quality of care
  Interventions: Behavioral: Ananya
- Control Condition (No Intervention): standard of care public health services in India

INTERVENTIONS:
Behavioral: Ananya — The Ananya program was developed and implemented via a partnership of the Bill and Melinda Gates Foundation and the Government of Bihar as a means of improving reproductive, maternal, newborn and child health (RMNCH) outcomes in the state, in particular focusing on improving health behaviors and service utilization in the final trimester of pregnancy and early postpartum period. Ananya was designed as a series of supply- and demand-side efforts to improve health. Efforts were focused on strengthening outreach services in quantity and quality, improving quality of facility services, and mobilizing communities to improve health behaviors. The Ananya program included training, mobilizing, and monitoring of government frontline health workers (FLWs, including anganwadi workers- AWWS, auxiliary nurse midwives- ANMs, and community health workers-ASHAs) to increase quantity and quality of home visits for RMNH screenings and services, and media messages to increase demand for services.
  Arms: Ananya Intervention

SUMMARY:
Ananya was funded by BMGF to reduce maternal, newborn, and child mortality; fertility; and child undernutrition in Bihar, India. Ananya involved multi-level interventions designed to build front line health worker (FLW) capacities and reach to communities and households, as well as to strengthen public health facilities and quality of care to increase maternal and neonatal care and health behaviors, and thus survival. From 2012 to 2014, eight focal districts in western and central Bihar.received Ananya, while 30 districts did not. Data were collected from mothers of infants 0-11 months at baseline and mothers of infants 0-23 months at 2 year follow-up, from comparable public health blocks in Ananya and Control districts to assess Ananya effects on quality and quantity of FLW home visits, postnatal health behaviors, and among older infants/toddlers, complementary feeding and vaccination. Difference in difference analyses were used to assess Ananya outcome effects in this quasi experimental study.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of infants 0-23 months residing in the catchment area of the subcenters (public health facilities) included in this study.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27633 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Receipt of two or more home visits from an FLW in the final trimester of pregnancy, using maternal survey response | 2 year follow up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months; item created for Ananya Survey
Receipt of any postnatal home visits from an FLW (in the first 24 hours at home after delivery and in first month following delivery), using maternal survey response | 2-year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months; items created for Ananya Survey
Postnatal care behaviors (4 outcomes)- clean cord care, KMC, delayed bath, initiation of breastfeeding), reported by mothers | 2 year follow-up
  Postnatal care practices [Nothing applied to cord or umbilicus; Health worker placed child unclothed on mother's chest/abdomen in skin-to-skin contact; First bath delayed by two or more days; Breastfed child within one hour of birth] assessed via self-report using a single item for each behavior from representative sample of mothers of children aged 0-11 months; items from demographic and health surveys
Any complementary feeding of solid or semisolid food for infants aged 6-11 months, using maternal survey response | 2 year follow-up
  a survey item was used to assesse complementary feeding of infants as reported by mothers of infants aged 0-11 months; items taken from the Demographic and Health Survey
Immunizations (4 outcomes)- receipt of DBT1 and DBT3 for infants 6-11 mo; receipt of DPT3 and measles vaccine for children 12-23 months, using immunization cards or maternal self report if not card | 2 year follow-up
  data from immunization cards or from self-reports when women did not have cards; approximately 50-60% of participants did not have immunization cards

CONTACTS AND LOCATIONS:
Overall Officials: Yamini Atmavilas, Principal Investigator — Bill and Melinda Gates Foundattion

IPD SHARING:
Plan to Share IPD: Yes
Data from this study are public and available from the Bill and Melinda Gates Foundation

REFERENCES:
- [Derived] Abdalla S, Pair E, Mehta K, Ward V, Mahapatra T, Darmstadt GL. Improving the precision of maternal, newborn, and child health impact through geospatial analysis of the association of contextual and programmatic factors with health trends in Bihar, India. J Glob Health. 2022 Nov 23;12:04064. doi: 10.7189/jogh.12.04064. PMID 36412069
- [Derived] Ward V, Abdalla S, Raheel H, Weng Y, Godfrey A, Dutt P, Mitra R, Sastry P, Chamberlain S, Shannon M, Mehta K, Bentley J, Darmstadt Md GL; Ananya Study Group. Implementing health communication tools at scale: mobile audio messaging and paper-based job aids for front-line workers providing community health education to mothers in Bihar, India. BMJ Glob Health. 2021 Jul;6(Suppl 5):e005538. doi: 10.1136/bmjgh-2021-005538. PMID 34312155
- [Derived] Darmstadt GL, Weng Y, Pepper KT, Ward VC, Mehta KM, Borkum E, Bentley J, Raheel H, Rangarajan A, Bhattacharya D, Tarigopula UK, Nanda P, Sridharan S, Rotz D, Carmichael SL, Abdalla S, Munar W; Ananya Study Group. Impact of the Ananya program on reproductive, maternal, newborn and child health and nutrition in Bihar, India: early results from a quasi-experimental study. J Glob Health. 2020 Dec;10(2):021002. doi: 10.7189/jogh.10.021002. Epub 2020 Dec 19. PMID 33427822
- [Derived] Abdalla S, Weng Y, Mehta KM, Mahapatra T, Srikantiah S, Shah H, Ward VC, Pepper KT, Bentley J, Carmichael SL, Creanga A, Wilhelm J, Tarigopula UK, Nanda P, Bhattacharya D, Atmavilas Y, Darmstadt GL; Ananya Study Group. Trends in reproductive, maternal, newborn and child health and nutrition indicators during five years of piloting and scaling-up of Ananya interventions in Bihar, India. J Glob Health. 2020 Dec;10(2):021003. doi: 10.7189/jogh.10.021003. PMID 33427818
- [Derived] Ward VC, Weng Y, Bentley J, Carmichael SL, Mehta KM, Mahmood W, Pepper KT, Abdalla S, Atmavilas Y, Mahapatra T, Srikantiah S, Borkum E, Rangarajan A, Sridharan S, Rotz D, Bhattacharya D, Nanda P, Tarigopula UK, Shah H, Darmstadt GL; Ananya Study Group. Evaluation of a large-scale reproductive, maternal, newborn and child health and nutrition program in Bihar, India, through an equity lens. J Glob Health. 2020 Dec;10(2):021011. doi: 10.7189/jogh.10.021011. Epub 2020 Dec 19. PMID 33425335
- [Derived] Ghosh R, Spindler H, Dyer J, Christmas A, Cohen SR, Das A, Sonthalia S, Mahapatra T, Gore A, Shah H, Walker DM. Simulation and team training embedded nurse mentoring programme and improvement in intrapartum and newborn care in a low-resource setting in Bihar, India. J Glob Health. 2020 Dec;10(2):021010. doi: 10.7189/jogh.10.021010. Epub 2020 Dec 19. PMID 33425334
- [Derived] Creanga AA, Jiwani S, Das A, Mahapatra T, Sonthalia S, Gore A, Kaul S, Srikantiah S, Galavotti C, Shah H. Using a mobile nurse mentoring and training program to address a health workforce capacity crisis in Bihar, India: Impact on essential intrapartum and newborn care practices. J Glob Health. 2020 Dec;10(2):021009. doi: 10.7189/jogh.10.021009. PMID 33425333
- [Derived] Mehta KM, Irani L, Chaudhuri I, Mahapatra T, Schooley J, Srikantiah S, Abdalla S, Ward V, Carmichael SL, Bentley J, Creanga A, Wilhelm J, Tarigopula UK, Bhattacharya D, Atmavilas Y, Nanda P, Weng Y, Pepper KT, Darmstadt GL; Ananya Study Group. Health layering of self-help groups: impacts on reproductive, maternal, newborn and child health and nutrition in Bihar, India. J Glob Health. 2020 Dec;10(2):021007. doi: 10.7189/jogh.10.021007. Epub 2020 Dec 19. PMID 33425331
- [Derived] Mehta KM, Irani L, Chaudhuri I, Mahapatra T, Schooley J, Srikantiah S, Abdalla S, Ward VC, Carmichael SL, Bentley J, Creanga A, Wilhelm J, Tarigopula UK, Bhattacharya D, Atmavilas Y, Nanda P, Weng Y, Pepper KT, Darmstadt GL; Ananya Study Group. Health impact of self-help groups scaled-up statewide in Bihar, India. J Glob Health. 2020 Dec;10(2):021006. doi: 10.7189/jogh.10.021006. Epub 2020 Dec 19. PMID 33425330
- [Derived] Ward VC, Raheel H, Weng Y, Mehta KM, Dutt P, Mitra R, Sastry P, Godfrey A, Shannon M, Chamberlain S, Kaimal R, Carmichael SL, Bentley J, Abdalla S, Pepper KT, Mahapatra T, Srikantiah S, Borkum E, Rangarajan A, Sridharan S, Rotz D, Nanda P, Tarigopula UK, Atmavilas Y, Bhattacharya D, Darmstadt GL; Ananya Study Group. Impact of mHealth interventions for reproductive, maternal, newborn and child health and nutrition at scale: BBC Media Action and the Ananya program in Bihar, India. J Glob Health. 2020 Dec;10(2):021005. doi: 10.7189/jogh.10.021005. Epub 2020 Dec 19. PMID 33425329
- [Derived] Abdalla S, Pair E, Mehta KM, Ward VC, Darmstadt GL. Geospatial variations in trends of reproductive, maternal, newborn and child health and nutrition indicators at block level in Bihar, India, during scale-up of Ananya program interventions. J Glob Health. 2020 Dec;10(2):021004. doi: 10.7189/jogh.10.021004. PMID 33425328